CLINICAL TRIAL: NCT06702124
Title: Effects of Dopaminergic Therapy in Patients with Alzheimer's Disease: a 24 Weeks Prospective, Randomized, Double-blind, Placebo-controlled, Parallel Group, International, Multi-center Phase III Study Evaluating Efficacy and Safety of Rotigotine 4 Mg/24 Hrs in Combination with Rivastigmine 9.5 Mg/24 Hrs in Mild to Moderate Alzheimer's Disease Patients.
Brief Title: A Phase 3 Study of Rotigotine in Combination with Rivastigmine in Mild to Moderate Alzheimer's Disease
Acronym: DOPAD-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU CT Number:2023-504602-11-00
Record Dates: First submitted 2024-11-12; First posted 2024-11-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
Keywords: Dopamine; Rotigotine
MeSH Terms: conditions — Alzheimer Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rotigotine 4 mg (Experimental): Rotigotine 4 mg/24 hours transdermal patch administration
  Interventions: Drug: Rotigotine 4Mg/24Hrs Patch
- Placebo (Placebo Comparator): Placebo transdermal patch administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine 4Mg/24Hrs Patch — Rotigotine 4 mg/24Hrs administration for 24 weeks
  Arms: Rotigotine 4 mg
Drug: Placebo — Placebo administration for 24 weeks
  Arms: Placebo

SUMMARY:
This is a 24-week prospective, randomized, double-blind, placebo-controlled, multi-center phase III study evaluating efficacy and safety of rotigotine 4mg/24 hrs in combination with rivastigmine 9.5 mg/24 hrs in mild to moderate AD patients. The total study duration per patient from baseline to the end will be 24 weeks. The study has a placebo-controlled design to eliminate experimental biases that arise from a participants' expectations, observer's effect on the participants, observer bias, confirmation bias, and other sources.

DETAILED DESCRIPTION:
Patients will be screened at trial sites for determination of eligibility to enter the study on the basis of diagnostic evaluations, according to current diagnostic criteria for probable AD, and safety assessments (vital sign complete physical and neurological examinations). The efficacy assessments (cognitive/behavioral evaluations) will be performed at Baseline before starting treatment and repeated ontreatment at Weeks 6, 12 and 24. EEG neurophysiological examinations will be performed at Baseline and at Week 24. Plasma biomarkers will be collected at baseline and at Week 24. Visit windows are ±7 days for all the scheduled visits. At each in-clinic visit (or upon early termination), AEs will be recorded, at screening, baseline, weeks 6, 12 and 24 vital signs measured, and physical and neurological examination performed. During intervening times between visits, caregivers will be contacted by telephone at approximately at Weeks 4 and 16 and an unscheduled visit will take place if needed in response to a safety concern.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-childbearing potential, as defined in Appendix 2) with a diagnosis of AD according to IWG criteria
2. Age 50-85 years
3. MRI or computerized tomography (CT) assessment, corroborating the clinical diagnosis of AD and excluding other potential causes of dementia, especially cerebrovascular lesions (see exclusion criteria, number 3)
4. Patients who show CSF biomarker data supporting the diagnosis of AD (for Czech Republic only: lumbar punctures can be performed for screening purposes), or patients with a positive Amyloid Pet Scan will qualify for the study
5. Stable on a treatment with rivastigmine transdermal patch for at least 3 months, of which at least the last month was at 9.5mg/day, or for one month, if the patient had received donepezil before rivastigmine
6. Mild to moderate stage of AD according to MMSE ≥18 and ≤26
7. Clinical Dementia Rating (CDR) total score of 0.5 or 1 (mild)
8. Evidence of frontal lobe dysfunctions as assessed by FAB ≤14
9. Absence of major depressive disease according to GDS of < 5
10. Formal education for five or more years
11. Previous decline in cognition for more than six months as documented in patient medical records
12. A caregiver available and living in the same household or interacting with the patient and available if necessary to assure administration of drug
13. Patients living at home or nursing home setting without continuous nursing care
14. General health status acceptable for a participation in a 6-month clinical trial
15. Stable pharmacological treatment of any other chronic condition for at least one month prior to screening
16. No regular intake of prohibited medications
17. Signed informed consent by the patient. If there are any doubts that the patient is mentally capable of giving informed consent, the patient will be examined and verified to be mentally capable by an independent physician/ neurologist, prior to the initiation of any study specific procedure. Signed consent of the caregiver

Exclusion Criteria:

1. Failure to perform screening or baseline examinations
2. Hospitalization or change of chronic concomitant medication one month prior to screening or during screening period
3. Clinical, laboratory or neuro-imaging findings consistent with:

   * other primary degenerative dementia (dementia with Lewy bodies, fronto- temporal dementia, Huntington's disease, Creutzfeldt-Jakob Disease, Down's syndrome, etc.);
   * other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.);
   * orthostatic hypotension and autonomic disorders
   * cerebrovascular disease (major infarct, one strategic or multiple lacunar infarcts, extensive white matter lesions > one quarter of the total white matter);
   * other central nervous system diseases (severe head trauma, tumors, subdural hematoma or other space occupying processes, etc.);
   * seizure disorder;
   * other infectious, metabolic, or systemic diseases affecting the central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, serum electrolytes out of normal range, juvenile onset diabetes mellitus, etc.).
4. A current DSM-V diagnosis of active major depression, schizophrenia, or bipolar disorder
5. Any suicidal ideation or suicidal behavior in the C-SSRS (C-SSRS score > 0)
6. Clinically significant, advanced, or unstable disease that may interfere with primary or secondary variable evaluations, and which may bias the assessment of the clinical or mental status of the patient or put the patient at special risk, such as:

   * history of any kind of psychosis
   * chronic liver disease, liver function test abnormalities or other signs of hepatic insufficiency (ALT, AST, Gamma GT, alkaline phosphatase > 2.5 ULN);
   * respiratory insufficiency;
   * renal insufficiency (serum creatinine >2 mg/dl) or creatinine clearance ≤ 30 mL/min according to Cockcroft-Gault formula). In case of creatinine clearance ≤30 mL/min, an alternative verification of the renal function must be completed using Cystatin C analysis. In case of normal level of Cystatin C, the patient can be included;
   * heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within six months before screening);
   * bradycardia (heart beat <50/min.) or tachycardia (heart beat >95/min);
   * hypertension (>140/90 mm/Hg) or hypotension (<90/60 mm/Hg) requiring treatment with more than three drugs;
   * AV block (type II / Mobitz II and type III), congenital long QT syndrome, sinus node dysfunction or prolonged QTcB-interval (males >450 and females >470 msec);
   * uncontrolled diabetes defined by HbA1c >8.5;
   * malignancies within the last five years except skin malignancies (other than melanoma) or indolent prostate cancer;
   * metastases;
   * disability that may prevent the patient from completing all study requirements (e.g. blindness, deafness, severe language difficulty, etc.);
   * women who are fertile and of childbearing potential;
   * chronic daily drug intake of ≥ 14 days or expected for ≥ 14 days:
   * benzodiazepines, neuroleptics or major sedatives,
   * antiepileptics,
   * centrally active anti-hypertensive drugs (clonidine, l-methyl DOPA, guanidine, guanfacine, etc.),
   * opioid containing analgesics,
   * nootropic drugs (except Ginkgo Biloba);
   * suspected or known drug or alcohol abuse, i.e., more than approximately 60 g alcohol (approximately 1 liter of beer or 500 ml of wine) per day, indicated by elevated mean corpuscular volume (MCV) above normal value at screening; (Please advise all subjects that because of possible additive effects, patients should not be taking alcohol in combination with rotigotine).
   * suspected or known allergy to any components of the study treatments;
   * hypersensitivity to the active substance rotigotine or to any of the excipients contained in the patches (according to SmPC).
   * enrollment in another investigational study or intake of investigational drug within the previous three months or five times the half-life of the IMP/metabolites (whichever is longer)
   * any condition, which, in the opinion of the investigator, makes the patient unsuitable for inclusion;
   * if the patient is in any way dependent on the sponsor or the principal investigator or if the patient is accommodated in an establishment on judicial or administrative order.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 24 in the FAB to evaluate efficacy of rotigotine in combination with rivastigmine on frontal lobe cognitive functions as compared to rivastigmine in combination with placebo. | From enrollment to the end of 24 weeks of treatment
  FAB is a brief battery of six neuropsychological tasks designed to assess frontal lobe function

SECONDARY OUTCOMES:
Change from Baseline to Week 24 in the ADCS-ADL to evaluate efficacy of rotigotine in combination with rivastigmine on autonomies of daily living as compared to rivastigmine in combination with placebo | From enrollment to the end of 24 weeks of treatment
  The ADCS-ADL includes 23 items that were derived from a larger set of items describing performance of activities of daily living
Change from Baseline to Week 24 in the MoCA to evaluate efficacy of rotigotine in combination with rivastigmine on cognition as compared to rivastigmine in combination with placebo. | From enrollment to the end of 24 weeks of treatment
  The MoCA is a brief, simple, and reliable screening test for AD. The test checks language, memory, visual and spatial thinking, reasoning, and orientation skills.
Change from Baseline to Week 24 in the CDR-SOB, to evaluate efficacy of rotigotine in combination with rivastigmine on cognition as compared to rivastigmine in combination with placebo | From enrollment to the end of 24 weeks of treatment
  The CDR is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to AD and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care
Change from Baseline to Week 24 in the ADAS-Cog14 to evaluate efficacy of rotigotine in combination with rivastigmine on memory functions as compared to rivastigmine in combination with placebo. | From enrollment to the end of 24 weeks of treatment
  ADAS-cog assesses the level of cognitive dysfunction in AD. The ADAS-Cog14 consists of items from the following areas chosen for their sensitivity to AD: language; memory; praxis executive functions and orientation.
Change from Baseline to Week 24 in the AMI to evaluate efficacy of rotigotine in combination with rivastigmine on levels of apathy and motivation as compared to rivastigmine in combination with placebo. | From enrollment to the end of 24 weeks of treatment
  The Apathy-Motivation Index was developed as a brief self-report index of apathy and motivation.

OTHER OUTCOMES:
Change from Baseline to Week 24 in the EEG recordings, to evaluate effects of rotigotine in combination with rivastigmine or rivastigmine in combination with placebo on cortical oscillatory activity. | From enrollment to the end of 24 weeks of treatment
  All patients will undergo resting EEG recordings at the beginning and at the end of the experimental protocol with a 21 channels EEG. The neurophysiological measurement will be performed with the eyes closed and will last 3 minutes.
Change from Baseline to Week 24 in plasma Neurofilament light chain (NfL) and Aβ42 and p-tau concentrations to evaluate effects of rotigotine in combination with rivastigmine in combination with placebo on plasma biomarkers | From enrollment to the end of 24 weeks of treatment
  Plasma samples will be collected according to the trail schedule

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Lucia Foundation, Rome, Italy, Italy